CLINICAL TRIAL: NCT02392676
Title: A Phase III, Randomised, Double Blind, Placebo Controlled, Multicentre Study of Olaparib Maintenance Monotherapy in Patients With Platinum Sensitive Relapsed Ovarian Cancer Who Are in Complete or Partial Response Following Platinum Based Chemotherapy and Whose Tumours Carry Loss of Function Somatic BRCA Mutation(s) or Loss of Function Mutation(s) in Tumour Homologous Recombination Repair -Associated Genes
Brief Title: Olaparib Maintenance Treatment Versus Placebo in Patients With PSR Ovarian Cancer Who Are in CR or PR to Platinum-based Chemotherapy and Whose Tumours Carry sBRCAm or HRR-associated Genes Mutations
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is unlikely to be feasible given the evolving ovarian cancer landscape and alternative studies have the potential to meet future clinical demand.
Sponsor: AstraZeneca (Industry)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D0816C00009
Record Dates: First submitted 2015-02-23; First posted 2015-03-19 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Platinum Sensitive Relapsed Ovarian Cancer
Keywords: Ovarian cancer; Platinum; Somatic BRCA mutation; Homologous recombination repair
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1/OLAPARIB (Experimental): olaparib 300 mg oral tablets; twice daily
  Interventions: Drug: OLAPARIB
- 2/PLACEBO (Placebo Comparator): placebo matching olaparib 300 mg oral tablets; twice daily
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: OLAPARIB — Patients should continue with therapy until objective radiological disease progression as per RECIST 1.1 despite rises in CA-125. All patients should continue to receive study treatment until objective radiological disease progression as per RECIST 1.1 as assessed by the investigator or the patient experiences unacceptable toxicity or they meet any other discontinuation criteria
  Arms: 1/OLAPARIB
Drug: PLACEBO — Patients should continue with therapy until objective radiological disease progression as per RECIST 1.1 despite rises in CA-125. All patients should continue to receive study treatment until objective radiological disease progression as per RECIST 1.1 as assessed by the investigator or the patient experiences unacceptable toxicity or they meet any other discontinuation criteria
  Arms: 2/PLACEBO

SUMMARY:
Olaparib administered as monotherapy in the maintenance setting improves progression free survival compared to placebo in patients whose tumours carry loss of function (deleterious or suspected deleterious) somatic BRCA mutations or loss of function (deleterious or suspected deleterious) mutation in non-BRCA Homologous Recombination Repair (HRR) -associated genes who have a complete or partial response to platinum-based chemotherapy.

DETAILED DESCRIPTION:
This is a phase III, randomised, double-blind, placebo-controlled, multi-centre study to assess the efficacy of olaparib maintenance monotherapy in relapsed high grade epithelial ovarian cancer patients (including patients with primary peritoneal and / or fallopian tube cancer) who have responded following platinum based chemotherapy. The study population will be enrolled as two separate cohorts that will enrol simultaneously. The confirmatory cohort will consist of patients who carry a somatic BRCA mutation (documented mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious) which are detected in tumour material but absent from germline blood testing ; the exploratory cohort will include patients with a mutation (documented mutation predicted to be deleterious or suspected deleterious) in non BRCA HRR-associated genes which are detected in tumour material regardless of their germline status.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age
* Histologically diagnosed relapsed high grade epithelial ovarian cancer (including primary peritoneal and/ or fallopian tube cancer)
* Documented deleterious or suspected deleterious somatic BRCA 1 and/or BRCA 2 somatic mutation or evidence of non- BRCA HRR-associated gene mutation in the tumour.
* At least 2 previous lines of platinum containing therapy prior to randomisation.
* CA-125 measurements prior to randomised treatment
* Patients must have normal organ and bone marrow function measured within 28 days of randomisation
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
* Provision of a blood sample for cfDNA biomarker analysis in Pre-Screening Part 1
* Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary or recurrent cancer must be available for central testing. If archival tumour sample is not available tumour sample from fresh biopsy is acceptable, for all patients eligible to participate in Pre-Screening part 2.

Exclusion Criteria:

* Documented germline mutation in BRCA1 and/or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function).
* Patients who have had drainage of their ascites from the final 2 cycles of their last chemotherapy regimen prior to randomisation on the study
* Participation in another clinical study with an investigational product during the chemotherapy course immediately prior to randomisation
* Any previous treatment with a PARP inhibitor, including olaparib
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product
* Prior malignancy in the last 5 years, unless curatively treated and recurrence free (few exceptions apply)
* Patients receiving any systemic chemotherapy (including chemotherapy received as the most recent anticancer therapy) or radiotherapy (except for palliative reasons) within 3 weeks prior to study randomised treatment
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) CTCAE grade 2) caused by previous cancer therapy, excluding CTCAE grade 2 peripheral neuropathy
* Patients with myelodysplastic syndrome/acute myeloid leukaemia (t-AML) or with features suggestive of MDS/AML
* Patients with symptomatic uncontrolled brain metastases
* Major surgery within 2 weeks of starting study randomised treatment and patients must have recovered from any effects of any major surgery
* Patients considered a poor medical risk

Ages: 18 Years to 96 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) using modified RECIST 1.1 in the cohort of patients with sBRCA ovarian cancer | From date of randomization until the date of first documented progression or date of death (by any cause, in the absence of disease progression) whichever came first, assessed up to 40 months
  To determine the efficacy of olaparib maintenance monotherapy compared to placebo by assessment of progression free survival (PFS) using blinded independent central review (BICR)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) using modified RECIST 1.1. in the Intent to Treat Population (ITT) consisting of all randomised patients with sBRCAm or HRR-associated gene mutations | From date of randomization until the date of first documented progression or date of death (by any cause, in the absence of disease progression), whichever came first, assessed up to 60 months
  To determine the efficacy of olaparib maintenance monotherapy compared to placebo by assessment of progression free survival (PFS)using blinded independent central review (BICR)
Overall Survival (OS) in patients with sBRCAm ovarian cancer and in the ITT population consisting of all randomised patients | From the date of randomisation until death due to any cause, assessed up to 60 months
  To determine the efficacy of olaparib maintenance monotherapy compared to placebo by assessment of overall survival (OS)
Time from randomisation to first subsequent therapy or death (TFST) in patients with sBRCAm ovarian cancer and in the ITT population consisting of all randomised patients | From the date of randomisation to the earlier of first subsequent therapy start date, assessed up to 60 months
  To determine the efficacy of olaparib maintenance monotherapy compared to placebo by assessment of Time from randomisation to first subsequent therapy or death
Trial outcome index (TOI) of the Functional Assessment of Cancer Therapy - Ovarian (FACT-O) in sBRCA and HRR associated gene mutated relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy | Administered at baseline, at day 29 then every 8 weeks (+/- 1 week) regardless of treatment discontinuation or disease progression, assessed up to 24 months
  To compare the effects of olaparib maintenance monotherapy compared to placebo on Health-related Quality of Life (HRQoL)
Plasma mutation status | cfDNA sample collected during pre-screening, assessed up to 40 months
  To determine if p53, somatic BRCA and other HRR mutations are present in plasma prior to chemotherapy
Time to earliest progression by RECIST 1.1 or CA-125 or Death in patients with sBRCAm ovarian cancer and in the ITT population consisting of all randomised patients | From randomisation to the earliest date of investigator assesed RECIST or CA-125 progression or death by any cause, assessed up to 60 months
  To determine the efficacy of olaparib maintenance monotherapy compared to placebo by assessment of Time to earliest progression by RECIST 1.1 or CA-125 or Death. Progression or recurrence based on serum CA-125 levels will be defined on the basis of a progressive serial elevation of serum CA-125
Time from randomisation to second progression (PFS2) in patients with sBRCAm ovarian cancer and in the ITT population consisting of all randomised patients | From the date of randomisation to the earliest of the progression event subsequent to that used for the primary variable PRS or death, assessed up to 60 months
  To determine the efficacy of olaparib maintenance monotherapy compared to placebo by assessment of Time from randomisation to second progression
Time from randomisation to second subsequent therapy or death (TSST) in patients with sBRCAm ovarian cancer and in the ITT population consisting of all randomised patients | From the date of randomisation to the earlier of the date of second subsequent chemotherapy start date or death date, assessed up to 60 months
  To determine the efficacy of olaparib maintenance monotherapy compared to placebo by assessment of Time from randomisation to second subsequent therapy of death
Time from randomisation to study treatment discontinuation or death (TDT) in patients with sBRCAm ovarian cancer and in the ITT population consisting of all randomised patients | From the date of randomisation to the earlier of the date of study treatment discontinuation or death, assessed up to 60 months
  To determine the efficacy of olaparib maintenance monotherapy compared to placebo by assessment of Time from randomisation to study treatment discontinuation or death

OTHER OUTCOMES:
Number of AEs in all patients who received at least one dose of randomised investigational product, olaparib or placebo | assessed up to 60 months
  To assess the safety and tolerability of olaparib maintenance monotherapy by assessment of AEs
Changes in Vital signs in all patients who received at least one dose of randomised investigational product, olaparib or placebo | assessed up to 60 months
  To assess the safety and tolerability of olaparib maintenance monotherapy by assessment of vital signs
Changes in Physical examination results in all patients who received at least one dose of randomised investigational product, olaparib or placebo | assessed up to 60 months
  To assess the safety and tolerability of olaparib maintenance monotherapy by assessment of physical examination parameters
Changes in safety laboratory parameters in all patients who received at least one dose of randomised investigational product, olaparib or placebo | assessed up to 60 months
  To assess the safety and tolerability of olaparib maintenance monotherapy by safety laboratory (consisting of clinical chemistry and haematology)parameters assessment

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Gourley, Prof., Principal Investigator — University of Edinburgh; Carol Aghajanian, MD, Principal Investigator — MSKCC
Locations (29):
- United States (15):
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Stanford, California
  - Research Site, Augusta, Georgia
  - Research Site, Park Ridge, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Albany, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Milwaukee, Wisconsin
- Peru (2):
  - Research Site, Chiclayo
  - Research Site, Lima
- Research Site, Quezon City, Philippines
- South Korea (3):
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Sutton